CLINICAL TRIAL: NCT05548114
Title: Randomized Trial Comparing Endoscopic Ultrasound-guided Gastrojejunostomy and Surgical Gastrojejunostomy in Gastric Outlet Obstruction
Brief Title: Randomized Trial of EUS-guided Gastrojejunostomy and Surgical Gastrojejunostomy in Gastric Outlet Obstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orlando Health, Inc. (Other)
Collaborators: West Virginia University (Other); Rush University (Other); Asian Institute of Gastroenterology, India (Other); Medanta, The Medicity, India (Other); University of Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22.127.06
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Gastric Outlet Obstruction
Keywords: Gastric outlet obstruction; Endoscopic ultrasound; Surgery; Malignancy; Gastrojejunostomy
MeSH Terms: conditions — Gastric Outlet Obstruction; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EUS-guided gastrojejunostomy (Active Comparator): EUS-guided gastrojejunostomy is performed using a lumen-apposing metal stent
  Interventions: Procedure: EUS-guided gastrojejunostomy
- Surgical gastrojejunostomy (Active Comparator): A surgical gastrojejunostomy will be created via laparoscopic or robotic techniques (preferred) or open technique (if these methods fail), as clinically appropriate.
  Interventions: Procedure: Surgical gastrojejunostomy

INTERVENTIONS:
Procedure: EUS-guided gastrojejunostomy — AXIOS lumen-apposing metal stent will be used to create a gastrojejunostomy under EUS guidance.
  Arms: EUS-guided gastrojejunostomy
Procedure: Surgical gastrojejunostomy — A surgical gastrojejunostomy will be created via laparoscopic or robotic techniques (preferred) or open technique (if these methods fail), as clinically appropriate.
  Arms: Surgical gastrojejunostomy

SUMMARY:
Malignant gastric outlet obstruction (GOO) results from the mechanical obstruction of the duodenum or distal stomach from an underlying cancer. The aim of this study is to compare the clinical outcomes between surgical gastrojejunostomy and EUS-guided gastrojejunostomy in patients with malignant gastric outlet obstruction.

DETAILED DESCRIPTION:
Malignant gastric outlet obstruction (GOO) results from the mechanical obstruction of the duodenum or distal stomach from an underlying cancer. The consequences of GOO are abdominal pain, nausea, vomiting, anorexia, inability to maintain an oral diet and weight loss, with associated poor quality of life and inability to continue with cancer therapy. The aim of this study is to compare the clinical outcomes between surgical gastrojejunostomy and EUS-guided gastrojejunostomy in patients with malignant gastric outlet obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Presence of gastric outlet or duodenal obstruction on any imaging or endoscopy from known or suspected inoperable malignancy
3. Gastric outlet obstruction Scoring System (GOOSS) of ≤ 1 (defined as maximum oral intake of liquids only)
4. Amenable to treatment by both EUS-guided and surgical gastrojejunostomy

Exclusion Criteria:

1. Age < 18 years
2. Intrauterine pregnancy
3. Use of anticoagulants that cannot be discontinued for the procedure or irreversible coagulopathy
4. Unable to obtain consent for the procedure from either the patient or LAR
5. Altered anatomy due to prior gastroduodenal surgery
6. Presence of other adhesions or synchronous obstructive lesions in the small bowel
7. Prior treatment for gastric outlet obstruction
8. Presence of large volume malignant ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite end point of inability to tolerate a solid diet (defined as gastric outlet obstruction scoring system score <2) or requiring additional interventions or supplemental nutrition or procedure-related adverse events. | 6 months
  Proportion of patients unable to tolerate a solid diet at time of hospital discharge (defined as gastric outlet obstruction scoring system score <2) or requiring additional interventions or supplemental nutrition or procedure-related adverse events.

SECONDARY OUTCOMES:
Gastric Outlet Obstruction Scoring System (GOOSS) score of ≥ 2 at 1-month post-procedure, without the need for repeat intervention or supplemental nutrition such as the use of enteric feeding tubes or total parenteral nutrition (TPN). | 6 months
  Proportion of patients with Gastric Outlet Obstruction Scoring System (GOOSS) score of ≥ 2 at 1-month post-procedure, without the need for repeat intervention or supplemental nutrition such as the use of enteric feeding tubes or total parenteral nutrition (TPN).
Gastric Outlet Obstruction Scoring System (GOOSS) score of ≥ 2 at 6-month post-procedure, without the need for repeat intervention or supplemental nutrition such as the use of enteric feeding tubes or total parenteral nutrition (TPN). | 6 months
  Proportion of patients with Gastric Outlet Obstruction Scoring System (GOOSS) score of ≥ 2 at 6-month post-procedure, without the need for repeat intervention or supplemental nutrition such as the use of enteric feeding tubes or total parenteral nutrition (TPN).
Rate of technical success | 24 hours
  Technical success is defined as the successful creation of a gastrojejunal anastomosis by the originally assigned method.
Procedure duration | 24 hours
  Procedure duration for EUS-guided and surgical gastrojejunostomy procedures
Time to diet advancement | 1 month
  Time to liquid diet (GOOSS score 1), soft solid diet (GOOSS score 2) and regular solid diet (GOOSS score 3).
Time to recurrence of obstructive symptoms | 6 months
  Recurrence of obstructive symptoms, defined as the recurrence of obstructive symptoms (GOOSS score ≤ 1) after achieving GOOSS ≥ 2 for at least 7 days at any time during follow-up.
Rate of persistence of symptoms | 6 months
  Persistent of obstructive symptoms, defined as continuing symptoms up to 2 weeks after index procedure.
Rate of reintervention | 6 months
  Reintervention, defined as need for repeat treatment for persistent or recurrent obstructive symptoms. Reintervention can be any endoscopic or surgical therapy.
Total number of readmissions | 6 months
  Total no. of readmissions due to disease-related symptoms or procedure-related events.
Rate of adverse events due to procedures performed | 6 months
  Procedure-related adverse events
Rate of adverse events due to underlying disease | 6 months
  Disease-related adverse events
Total length of hospital stay | 6 months
  Duration of hospitalization, defined as the length of hospital stay from the date of the procedure to the date of discharge.
Length of survival | 6 months
  Duration of survival post-procedure.
Time to initiation of chemotherapy post-procedure | 6 months
  Time to initiation of chemotherapy post-procedure
Quality of life measurement | 6 months
  Quality of life post-procedure as determined by the EORTC-QLQ-C30 quality of life questionnaire.
Treatment costs | 6 months
  All relevant costs pertaining to treatment of gastric outlet obstruction will be taken into consideration from index intervention to hospital discharge: procedure costs, inpatient hospital stay from date of procedure to discharge, medications, materials, anesthesia, pharmacy and imaging studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bang JY, Puri R, Lakhtakia S, Thakkar S, Waxman I, Siddiqui I, Arnold K, Chaudhary A, Mehta S, Singh A, Venkat Rao G, Basha J, Gupta R, Modak S, Singh S, Boone B, Dautel P, Dixon MEB, Kim HM, Sutton B, Arnoletti JP, Rosch T, Varadarajulu S. Endoscopic or surgical gastroenterostomy for malignant gastric outlet obstruction: a randomised trial. Gut. 2025 Dec 5;75(1):24-32. doi: 10.1136/gutjnl-2025-336339. PMID 40998416